CLINICAL TRIAL: NCT01485705
Title: Frequency, Consequences and Determinants of Sub-optimal Care in the Initial Care of Severe Bacterial Infections of the Child
Brief Title: Retrospective Examination of Initial Care of Severe Bacterial Infections of the Child
Acronym: Diabact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BRD/08/06-T
Record Dates: First submitted 2011-09-06; First posted 2011-12-05 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Bacterial Infection
Keywords: severe bacterial infection
MeSH Terms: conditions — Bacterial Infections | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Retrospective examination by experts whether care given fo child admitted at the ICU for suspicion of bacterial infection (not nosocomial) was optimal or not — When child is admitted at Intensive Care Unit (ICU) for suspicion of bacterial infection that is not nosocomial, data on child's infection and cares received, is completed on an electronic Case Report Form (e-CRF) by Doctor of ICU. Characteristic "optimal or not" of initial medical care is then determined by the independent experts blinded from issue of the care.

SUMMARY:
The aim of the study is to determine the frequency of sub-optimal care in the initial care (before arrival at the intensive care unit) of children from "West France regions" suffering of severe bacterial infections.The characteristic "optimal or not" of the initial medical care will be determined by 2 independent experts, blinded from each other and blinded from the issue of the care. In case of a discordance between the two experts, a third expert will be demanded. Three possibilities of conclusion will be proposed to the experts: "sure sub-optimal medical care", "possible suboptimal care" and "optimal care".

ELIGIBILITY:
Inclusion Criteria:

* Child from West France regions
* Aged between 1 month and 16 years old,
* Admitted at the intensive care unit for a severe bacterial infection and with the first symptoms appeared when child was at home or hospitalized since less than 48h
* Children dead at home will also be included in this study via the mobil medical urgency help unit (french term : "SAMU")

Exclusion Criteria:

* Patient not fulfilling inclusion criteria
* Child with a nosocomial infection
* Child dead or admitted at the intensive care unit following a pertussis- Child not admitted at the intensive care or not dead at home in a context of infection.
* Child with viral or fungic infection admitted at the intensive care unit.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 371 (Actual)
Dates: Start 2009-08-13 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Frequency of optimal care and of non optimal care in the initial care (before arrival at the intensive care unit) of children (from West France regions) suffering of severe bacterial infections. | 1day
  For each child medical file, the verdict "optimal care" or the verdict " non optimal care" will be determined by two independent experts, blinded from each other. If verdict base their judgement through recommendations listed in the literature.

SECONDARY OUTCOMES:
characteristics of sub-optimal cares | 1 day
  Experts will explain their verdict by answering to a list of questions. These questions will allow to identify and classify characteristics of defaults of cares .
determinants of sub-optimal cares | 1 day
  To identify determinants of sub-optimal cares (examples : place of medical care, qualification and experience of the Medical Doctor, moment of medical care.
consequences of initial sub-optimal cares | 1 day
  To identify consequences of initial sub-optimal cares on the outcome of children with severe bacterial infections (child death, etc).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Nantes, Nantes, France

REFERENCES:
- [Derived] Malorey D, Lorton F, Chalumeau M, Bourgoin P, Boussicault G, Chantreuil J, Gaillot T, Roue JM, Martinot A, Assathiany R, Saulnier JP, Caillon J, Grain A, Gras-Le Guen C, Launay E. Distribution, Consequences, and Determinants of Time to Antibiotics in Children With Community-Onset Severe Bacterial Infection: A Secondary Analysis of a Prospective Population-Based Study. Pediatr Crit Care Med. 2023 Sep 1;24(9):e441-e451. doi: 10.1097/PCC.0000000000003306. Epub 2023 Jun 1. PMID 37260312